CLINICAL TRIAL: NCT01595724
Title: Study to Characterize Patients Treated With Visanne for Their Endometriosis Under Real-life Practice Conditions and Evaluate Their Quality of Life at Baseline and After 6 Months of Treatment With Visanne.
Brief Title: Daily Practice Treatment and Influence of Visanne on the Patient Assessment of Quality of Life
Acronym: DIVA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16108; VS1101 (Other: company internal)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Endometriosis
Keywords: Non-interventional study; Endometriosis,; Quality of life
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Visanne (Dienogest, BAY86-5258)

INTERVENTIONS:
Drug: Visanne (Dienogest, BAY86-5258) — Intake of Dienogest 2mg/day to treat Endometriosis according to regular clinical practice.

SUMMARY:
The study aims to collect data on the influence of a treatment with Visanne (Dienogest 2mg/d) on the Endometriosis related quality of life. These data will be collected using a special patient questionnaire (Endometriosis Health Profile 5, EHP-5). The study will also be used to describe the basic disease status and demographic characteristics of patients searching treatment by a gynecologist because of their endometriosis. In addition, the study will give insight into the typical diagnostic measures the physicians in different countries are using in the field of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 18 years of age
* Clinical or laparoscopic diagnosis of endometriosis
* Having endometriosis related pain as leading symptom
* Decision taken by physician to prescribe Visanne
* Signed Informed Consent Form

Exclusion Criteria:

* Contraindications listed in the local summary of product characteristics (SPC) have to be considered.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gynecological patients
Sampling Method: Probability Sample
Enrollment: 3006 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients, who show an improvement of the EHP-5 items | after 6 months of treatment
Mean changes of EHP-5 items by using scores for pre-defined categories | after 6 months of treatment

SECONDARY OUTCOMES:
Baseline demographic characteristics and disease status of patients with endometriosis treated with Visanne | Baseline
Patient reported severity of endometriosis related pain | Baseline and after 6 months of treatment
Reasons for treatment discontinuation | after 6 months of treatment
Safety variables will be summarized using descriptive statistics based on adverse events collection | after 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Many Locations, Belarus
- Many Locations, Egypt
- Many Locations, Jordan
- Many Locations, Kazakhstan
- Many Locations, Kuwait
- Many Locations, Lebanon
- Many Locations, Qatar
- Many Locations, Russia
- Many Locations, Saudi Arabia
- Many Locations, Ukraine
- Many Locations, United Arab Emirates